CLINICAL TRIAL: NCT06331221
Title: Effects of Different Concentric and Eccentric Muscle Fatigue Protocols on the Knee Joint Position Sense: a Randomized Controlled Crossover Trial
Brief Title: Effects of Different Concentric and Eccentric Muscle Fatigue Protocols on the Knee Joint Position Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: JSA_Fatigue_FADEUP
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Muscle Fatigue; Knee; Joint Position Sense; Proprioception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control Condition (No Intervention): 5-minute rest period.
- Quadriceps_Concentric (Active Comparator): 40 consecutive maximal concentric contractions of quadriceps at 30º/s
  Interventions: Other: Muscle fatigue Protocol
- Quadriceps_Eccentric (Active Comparator): 40 consecutive maximal eccentric contractions of quadriceps at 30°/s
  Interventions: Other: Muscle fatigue Protocol
- Hamstrings_Concentric (Active Comparator): 30 consecutive maximal concentric contractions of hamstrings at 30º/s
  Interventions: Other: Muscle fatigue Protocol
- Hamstrings_Eccentric (Active Comparator): 30 consecutive maximal eccentric contractions of the hamstrings at 30º/s
  Interventions: Other: Muscle fatigue Protocol

INTERVENTIONS:
Other: Muscle fatigue Protocol — Four experimental conditions consisting of different local muscle fatigue protocols performed in the isokinetic dynamometer in random order, with at least one week of interval between them.
  Arms: Hamstrings_Concentric; Hamstrings_Eccentric; Quadriceps_Concentric; Quadriceps_Eccentric

SUMMARY:
The aim of this study was to investigate the effects of different concentric and eccentric muscle fatigue protocols on the knee joint position sense of healthy individuals.

DETAILED DESCRIPTION:
A randomized controlled crossover trial will be conducted at a biomechanics laboratory with healthy males. All participants will perform with a washout period of 1 week: a control condition (5-minute rest) and 4 local muscle fatigue protocols (concentric of quadriceps; concentric of hamstrings; eccentric of quadriceps; eccentric of hamstrings) in an isokinetic dynamometer at 30º/s. Three maximum voluntary isometric contractions (MVIC) of quadriceps and hamstrings will also be assessed in the beginning of all conditions.

Knee joint position sense will be assessed before and immediately after the fatigue protocols/control condition, through active concentric and eccentric positionings/repositionings, in sitting and prone positions, to a target range of 45º of knee flexion in an isokinetic dynamometer. Surface electromyography electrodes will also be placed on the vastus lateralis and biceps femoris during all procedures.

ELIGIBILITY:
Inclusion Criteria:

* males aged between 18 and 30 years;
* without current or previous knee pathology or surgery;
* with a low or moderate physical activity level, according to the International Physical Activity Questionnaire;
* normal Body Mass Index (under 24.9 kg/m2), according to the World Health Organization.

Exclusion Criteria:

* those with cardiorespiratory, neurological or vestibular pathologies;
* with positive knee integrity tests (anterior drawer, Lachman's test, posterior drawer; valgus and varus stress testes); and
* those taking any medication that can affect motor control (sedatives, anxiolytics, antibiotics, analgesics, NSAIDs or myorelaxants).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Absolute angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The absolute value of the difference between the target range and the achieved range
Relative angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The arithmetic difference between the target range and the range achieved
Variable angular error | Change from Baseline (Before) to Immediately after interventions or control (After)
  The standard deviation of the 3 repositionings

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Desporto, Universidade do Porto, Porto, Portugal